CLINICAL TRIAL: NCT02977416
Title: Oxidation Rates of the Different Substrates During Exercise in Children and Adolescents With Juvenile Idiopathic Arthritis. Case-control Study and Cases Treated / Cases Not Treated With Anti-TNFα
Acronym: OSE-JIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: CHU-0295; 2016-A01262-49 (Other: 2016-A01262-49)
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Juvenile idiopathic arthritis; fat oxidation; exercise
MeSH Terms: conditions — Arthritis, Juvenile; Motor Activity

ARMS (3):
- patients treated withTNF blockade (Experimental): 22 patients treated with TNF blockade
  Interventions: Other: anti-TNFα
- patients without TNF blockade (Experimental): 22 patients without TNF blockade
  Interventions: Other: anti-TNFα
- healthy subjects (Experimental): 22 matched healthy subjects by pubertal stage and sex
  Interventions: Other: anti-TNFα

INTERVENTIONS:
Other: anti-TNFα

SUMMARY:
During exercise, energy comes mainly from carbohydrates and lipids. The relative contribution of lipids and glucose as energy substrates to exercise depends on the parameters of the exercise (duration, intensity and level of training) and the physiological conditions of the subject.

Inflammatory diseases such as juvenile idiopathic arthritis (JIA) are treated, for the most severe forms, by biotherapies. These treatments target certain pro-inflammatory cytokines including TNFα. In adults with rheumatoid arthritis several studies have shown that treatment with anti-TNFα increases insulin sensitivity. There is no data on the oxidation of energy substrates during exercise in children and adolescents with AJI, nor on the impact of anti-TNFα treatments on the oxidation of energetic substrates in children.

Investigators hypothesize that, compared to healthy children, children with JIA should exhibit altered oxidation of energy substrates at rest and submaximal physical exercise due to physical deconditioning and inflammation. In addition, those treated with anti-TNFα should have an oxidation profile of energy substrates at exercise different from that of patients not treated with anti-TNFα. Investigators also hypothesize that anti-TNFα treatments modify the contribution of energy chains (aerobic, anaerobic and anaerobic alactic) during the exercise.

DETAILED DESCRIPTION:
Annual evaluation by Lipoxmax test and Wingate anaerobic test (WAnT) during 3 years or until the transition from pediatric to adult care.

For healthy volunteer, only one lipaxmax and Wingate test.

ELIGIBILITY:
Inclusion Criteria:

* Children with juvenile idiopathic arthritis

Exclusion Criteria:

* active infection
* BMI > 25
* Systemic corticosteroid within last 3 months

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-05 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Percentage variation of the maximal fat oxidative rate during an exercise between JIA and healthy children. Timing: | at day 1 (first test)

SECONDARY OUTCOMES:
Percentage variation of substrates oxidative crossing point during an exercise. | at day 1
Description of the contribution of energy systems during supra-maximal physical exercise | at day 1 (first test)
  Description of the contribution of energy systems during supra-maximal physical exercise in patients with JIA according to JIA subtype, treatments, age, pubertal status, disease status

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermon-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Rochette E, Bourdier P, Pereira B, Dore E, Birat A, Ratel S, Echaubard S, Duche P, Merlin E. TNF blockade contributes to restore lipid oxidation during exercise in children with juvenile idiopathic arthritis. Pediatr Rheumatol Online J. 2019 Jul 22;17(1):47. doi: 10.1186/s12969-019-0354-1. PMID 31331342